CLINICAL TRIAL: NCT03121872
Title: Effectiveness and Predictability of Titanium-Prepared Platelet-Rich Fibrin for the Management of Multiple Gingival Recessions
Brief Title: Titanium Prepared Platelet Rich Fibrin for Multiple Gingival Recessions
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Karadeniz Technical University (Other)
Responsible Party: Principal Investigator, Esra Ercan, Asistant Proffesor Doctor, Karadeniz Technical University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2014/21; date: 07.04.2014
Record Dates: First submitted 2017-04-05; First posted 2017-04-20 (Actual); Last update posted 2017-04-24 (Actual); Status verified 2017-04

CONDITIONS: Gingival Recession
MeSH Terms: conditions — Gingival Recession

STUDY DESIGN:
Intervention Model Description: In this randomized controlled clinical trial, multiple gingival recessions were treated by T-PRF in 16 patients and by CTG in 18 patients selected by the coin-toss method. All surgical procedures, measurements and follow-up were performed by the same clinician
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Root Coverage Surgery with T-PRF (Experimental): Multiple gingival recessions were treated by Titanium prepared PRF (T-PRF) in 16 patients.
  The T-PRF membrane that was procured was placed in the defect area 1 mm beyond the enamel-cement border.. The T-PRF was fixed in the receiver area by a mattress stitch through the apical aspect using 5-0 monofilament absorbable sutures. The flap was stitched in a manner that completely covered the graft in the coronal aspect. Thereafter, the graft was fixed to the flap on the coronal aspect with horizontal mattress sutures. Compression was applied to the receiver area with serum-impregnated sterile gauze for approximately 5 minutes, and then periodontal paste was placed onto the surgery site.
  Interventions: Procedure: Root Coverage Surgery with T-PRF
- Root Coverage Surgery with CTG (Active Comparator): Multiple gingival recessions were treated by Connective Tissue Graft (CTG)in 18 patients.The CTG width was measured to include 1 mm beyond the root surface defects in the receiver area. Following anaesthesia of the palate, the borders of the start and finish incisions were marked. Subepithelial connective tissue that was 1.5-2 mm thick and excluded the periosteum was removed and maintained in physiological saline. The palate was stitched with 4-0 absorbable sutures (Pegalak, Doğsan, Turkey) and covered with a periodontal paste.
  Before placing the connective tissue in the receiver area, the fat and glandular tissues and the band-shaped epithelium on the connective tissue were removed using scissors.
  Interventions: Procedure: Root Coverage Surgery with CTG

INTERVENTIONS:
Procedure: Root Coverage Surgery with T-PRF — Root surfaces in the multiple gingival recession regions were made smooth using Gracey curettes. To remove the smear layer, 24% EDTA solution was applied to the tooth surfaces for approximately 2 minutes and then washed with physiological saline. The receiver region was prepared using the modified tunnel method. After passive stabilization of the flap in the coronal aspect, the preparation of the donor region was initiated
  Arms: Root Coverage Surgery with T-PRF
Procedure: Root Coverage Surgery with CTG — Root surfaces in the multiple gingival recession regions were made smooth using Gracey curettes. To remove the smear layer, 24% EDTA solution was applied to the tooth surfaces for approximately 2 minutes and then washed with physiological saline. The receiver region was prepared using the modified tunnel method. After passive stabilization of the flap in the coronal aspect, the preparation of the donor region was initiated
  Arms: Root Coverage Surgery with CTG

SUMMARY:
Objective: Titanium-prepared platelet-rich fibrin (T-PRF) is activated with titanium, which results in a more mature and aggregated form than PRF. In our previous studies, we established that the fibrin carpet formed with titanium had a firmer network structure, and longer resorption time in the tissue than the fibrin carpet formed with glass. The purpose of this randomized controlled clinical trial is to compare the effects of autogenous T-PRF and CTG.

Materials and methods: A total 114 Miller Class I/II gingival recessions with abrasion defects will be treated either T-PRF (63 teeth) or CTG (51 teeth) using a modified tunnel technique. Clinical periodontal indexes, keratinized tissue (KTW), gingival thickness (GT) and recession depth (RD) will be recorded before surgery and at 6 and 12-month follow-up examinations. The Visual Analog Scale and healing index scores will be assessed.

DETAILED DESCRIPTION:
A total of 34 patients will be informed in detail about the risks and benefits of each step of the study, and their signed consents will be obtained.

These clinical assessments will be done:

1. Plaque Index and Gingival Index In case of multiple gingival recessions, plaque index and gingival index will be obtained from the three dental points as mesial, distal and vestibule midpoints; plaque index will be calculated according to Sillnes&Löe criteria, whereas gingival index will be calculated according to Löe&Silness criteria.
2. Periodontal Pocket Depth In case of multiple gingival recessions, the distance between the pocket base and free gingival margin will be measured separately for each tooth with the assistance of periodontal Williams probe through the midpoint of vestibule.
3. Recession Width Periodontal probe will be horizontally placed on the enamel-cement border and the measurement will be recorded.
4. Recession Depth The defect distance will be measured vertically from the enamel-cement conjunction of the tooth to the very apical aspect of the gingival margin using periodontal probe and recorded in millimeters.
5. Clinical Attachment Level The clinical attachment level (CAL) will be measured by periodontal probe through the midpoint of vestibule as the distance between gingiva base and enamel-cement border and recorded in millimeters.
6. Keratinized Tissue Width The distance between gingival margin and alveolar mucosa will be measured in millimeters. A solution consisted of 10% potassium iodide and 5% iodine will be applied onto the gingiva and alveolar mucosa with a cotton pellet. This solution stains the glycogen-rich alveolar mucosa darker than the keratinized tissue and allows keratinized gingival mucosa to be exposed more clearly.
7. Gingival Thickness This measurement will be performed in the relevant area by No. 15 endodontic spreader under topical anesthesia. The spreader will be placed perpendicular to the gingiva through approximately 1.5 mm apical aspect of the gingival margin, pushed forward until obtaining bone support, and fixed with a disc. The distance between the disc and the tip of endochuck will be measured by a digital caliper with a sensitivity of 0.1 mm.
8. Measurement of CTG Thickness Fat and glandular tissue and band-shape epithelium on the CTG, which will be derived from the maxillary palate, will be removed by a scissor. The graft, which will be placed onto a sterile, metal smooth surface, will be fixed through its mesial, distal and middle aspects by a No. 15 endodontic spreader with the assistance of a disc and then measured by digital caliper. The mean graft thickness will be calculated as the arithmetic mean of the values measured.
9. Measurement of T-TRF Membrane Thickness Two thrombocyte rich platelets taken from the tubes that have been centrifuged will be separated from the serum at room temperature in sterile gauze and will be turned into membranes. They will be measured by digital caliper as two-layer similar to the measurement of connective tissue thickness, and the values will be recorded..

VAS Assessment On the postoperative Day 1, 3 and 7, the patients will be asked to complete a chart where they can rate subjective complaints of pain, burning sensation and discomfort in the surgery site between 0 (none) and 100 (very severe).

Wound Healing Index While removing the sutures two weeks after surgery, the physician will evaluate wound healing according to the Huang criteria separately for each tooth; Score 1: Problem-free wound healing without gingival edema, erythema, suppuration, or dehiscence of the flap margins.

Score 2. Problem-free wound healing with mild gingival edema, erythema, patient discomfort and flap dehiscence without suppuration.

Score 3. Poor wound healing with severe gingival edema, erythema, suppuration, patient discomfort and flap dehiscence.

Calculation of Root Surface Coverage Ratio This ratio is presented as percentage (%) and evaluated in the 6th and 12th months.

Preoperative recession depth - Postoperative recession depth X 100 % Preoperative recession depth

ELIGIBILITY:
Inclusion Criteria:

Eligibility criteria included the following:

* Absence of systemic disease that would likely hinder periodontal surgery or unfavourably influence wound healing
* Having multiple gingival recessions including at least two adjacent Miller class I or II teeth among mandibular or maxillary incisors and premolars. Molars were excluded.
* The teeth undergoing treatment were vital with no restoration or decay in the tooth neck (collum dentis) and with a completely or partially fixable enamel-cement border
* The relevant teeth in the arch were rotation-free with no mobility
* The presence of periodontal pockets not exceeding 3 mm in the teeth undergoing treatment; the teeth had no occlusal trauma; and the patients were older than 18 years of age

Exclusion Criteria:

* Receiving medicines that would likely cause gingival hypertrophy
* Smokers
* Presence of blood-borne diseases
* Presence of any systemic disease likely to influence coagulation, and receiving any anticoagulant medicines

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2014-05-21 (Actual); Primary Completion 2016-05-20 (Actual); Study Completion 2016-08-05 (Actual)

PRIMARY OUTCOMES:
Root Coverage Percentage at 12 months | Change from baseline Root Coverage Percentage at 12 months
  Preoperative recession depth - Postoperative recession depth X 100 % Preoperative recession depth

SECONDARY OUTCOMES:
Keratinized Tissue Width at 12 months | Change from baseline Keratinized Tissue Width at 12 months
  The distance between gingival margin to mucogingival junction

CONTACTS AND LOCATIONS:
Overall Officials: Esra Ercan, Study Director — Karadeniz Technical University
Locations (1):
- Esra Ercan, Trabzon, Others, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No